CLINICAL TRIAL: NCT06703463
Title: A Phase 1, Open-Label, Fixed-Sequence Study to Evaluate the Effect of Multiple Doses of Diltiazem on the Single-Dose Pharmacokinetics of MK-1167 in Healthy Adult Participants
Brief Title: A Drug-Drug Interaction Study of Diltiazem and MK-1167 in Healthy Adult Participants (MK-1167-006)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 1167-006; MK-1167-006 (Other: MSD)
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-1167 Period 1 (Experimental): On Day 1 a single dose of MK-1167 will be administered.
  Interventions: Drug: MK-1167
- MK-1167 Period 2 (Experimental): There will be a washout of at least 35 days between MK-1167 dosing in Period 1 and the first diltiazem dose in Period 2. In Period 2, diltiazem will be administered once daily (QD) for 49 consecutive days with a single dose of MK-1167 coadministered on Day 3.
  Interventions: Drug: MK-1167; Drug: Diltiazem

INTERVENTIONS:
Drug: MK-1167 — Administered via oral capsule per dosing regimen.
Drug: Diltiazem — Diltiazem hydrochloride administered at a dose of 240 mg QD via oral capsules.
  Arms: MK-1167 Period 2

SUMMARY:
The goal of this study this study is to learn about the safety of MK-1167 and if people tolerate it. Researchers will compare what happens to MK-1167 in the body when it is given with and without another medicine called diltiazem.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing based on participant self-reporting
* Body mass index (BMI) ≥18.0 and ≤32.0 kg/m^2
* Able to swallow multiple capsules
* In good health

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History or presence of second- or third-degree atrioventricular heart block (except in participants with a functional artificial pacemaker)
* History or presence of clinically significant sick sinus syndrome
* History of cancer (malignancy) within the past 5 years
* Unable to refrain from or anticipates the use of any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Number of participants who experience one or more adverse events (AEs) | Up to approximately 99 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study intervention due to an AE | Up to approximately 85 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Area under the concentration versus time curve from 0 to infinity after single dosing (AUC0-inf) of MK-1167 in plasma | Predose, and at designated timepoints up to 50 days post-dose
  AUC0-inf of MK-1167 in plasma will be determined.

SECONDARY OUTCOMES:
Area under the concentration versus time curve from 0 to last quantifiable sample (AUC0-last) of MK-1167 in plasma | Predose, and at designated timepoints up to 50 days post-dose
  AUC0-last of MK-1167 in plasma will be determined.
Maximum concentration (Cmax) of MK-1167 in plasma | Predose, and at designated timepoints up to 50 days post-dose
  Cmax of MK-1167 in plasma will be determined.
Concentration at hour 24 (C24) of MK-1167 in plasma | Predose, and at designated timepoints up to 24 hours post-dose
  C24 of MK-1167 in plasma will be determined.
Time to maximum concentration (Tmax) of MK-1167 in plasma | Predose, and at designated timepoints up to 50 days post-dose
  Tmax of MK-1167 in plasma will be determined.
Apparent terminal half-life (t1/2) of MK-1167 in plasma | Predose, and at designated timepoints up to 50 days post-dose
  t1/2 of MK-1167 in plasma will be determined.
Apparent clearance (CL/F) of MK-1167 in plasma | Predose, and at designated timepoints up to 50 days post-dose
  CL/F of MK-1167 in plasma will be determined.
Apparent volume of distribution during terminal phase (Vz/F) of MK-1167 in plasma | Predose, and at designated timepoints up to 50 days post-dose
  Vz/F of MK-1167 in plasma will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0002), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com